CLINICAL TRIAL: NCT06282120
Title: Efficacy and Safety of Irinotecan Liposome Injection Combined With 5-FU/LV± Immunotherapy in First-line Gemsitabine + Immunoprogressive Patients With Metastatic Biliary Tract Cancer
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSPC-DNY-BTC
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Arms: Drug: Irinotecan Hydrochloride Liposome Injection The recommended dose and regimen of Irinotecan Hydrochloride Liposome Injection is 70 mg/m2 intravenously over 90 minutes, followed by dl-LV 400mg/m2 or l-LV 200mg/m2 intravenously over 30 minutes, followed by 5-FU 2400 mg/m2 intravenously over 46 hours, administered every 3 weeks.It can be combined or partially combined immunotherapy.
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection ；Fluorouracil ；Leucovorin；immunotherapy

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection ；Fluorouracil ；Leucovorin；immunotherapy — The recommended dose and regimen of Irinotecan Hydrochloride Liposome Injection is 70 mg/m2 intravenously over 90 minutes, followed by dl-LV 400mg/m2 or l-LV 200mg/m2 intravenously over 30 minutes, followed by 5-FU 2400 mg/m2 intravenously over 46 hours, administered every 3 weeks.It can be combined or partially combined immunotherapy.
  Other Names: Liposomal irinotecan; 5-FU/LV

SUMMARY:
The goal of this clinical trial is to test in biliary tract cancer patients . The main questions it aims to answer are:

* To evaluate the efficacy of irinotecan liposome injection combined with 5-FU/LV± immunotherapy for first-line gemsitabine + immunoprogressive metastatic biliary tract cancer
* To evaluate the safety of irinotecan liposome injection combined with 5-FU/LV± immunotherapy for first-line gemsitabine + immunoprogressive metastatic biliary tract cancer This study intends to use liposomal irinotecan combined with 5-FU/LV± immunotherapy for second-line treatment of advanced biliary tract cancer that has progressed after gemsitabine + immunotherapy to evaluate the efficacy and safety of this regimen, with a view to providing better treatment options for second-line patients with advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patient had good compliance, could understand the research process of the study, and signed a written informed consent;
2. Age ≥18 years, ≤75 years;
3. Histologically or cytologically confirmed cholangiocarcinoma;
4. Documented metastatic disease;
5. At least one measurable lesion according to RECIST v1.1;
6. Disease progression after gemcitabine + immunotherapy;
7. For patients whose disease recurred after curative resection (R0 or R1), previous adjuvant 5-FU-based chemotherapy is allowed if there is at least 6 month-interval between the last dose of adjuvant chemotherapy and recurrence of disease;
8. Eastern Cooperative Oncology Group (ECOG) Performance status 0-1;
9. The expected survival time is greater than 3 months;
10. Having adequate organ function, as defined below:

    1. Absolute neutrophil count (ANC) ≥1.5*109/L
    2. Hemoglobin ≥90g/dL
    3. Platelets (PLT) ≥100*109/L
    4. Total bilirubin < 1.5 times Upper Normal Value (ULN)
    5. Chemical examination of liver function index (AST&ALT) < 2.5 times Upper Limit of Normal (ULN)
    6. Serum creatinine (Cr) ≤1.5×ULN
11. Non-pregnant or lactating women; Effective contraception should be used by women/men of childbearing age during the study period and for 6 months after the end of study treatment-

Exclusion Criteria:

（1) Serum total bilirubin ≥2 x ULN (upper limit of normal) (biliary obstruction allows biliary drainage); （2）Severe renal impairment (Clcr ≤ 30 ml/min); （3）Any clinically significant disorder impacting the risk-benefit balance negatively per physician's judgment； （4）Any clinically significant gastrointestinal disorder, including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 2; （5）Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) in last 6 months; （6） NYHA(New York Heart Association) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure. Or known abnormal ECG with clinically significant abnormal findings; （7） Active infection or an unexplained fever >38.5°C (excluding tumor fever), which in the physician's opinion might compromise the patient's health; （8） Current use or any use in last two weeks of strong CYP3A-enzyme inducers/inhibitors and/or strong UGT1A inhibitors； （9） Known hypersensitivity to any of the components of Onivyde other liposomal irinotecan formulations, irinotecan, fluoropyrimidines, or leucovorin; （10）Breast feeding, known pregnancy, positive serum pregnancy test or unwillingness to use an effective method of contraception, during therapy and for 3 months following the last dose of Onivyde. Females of Childbearing Potential must either agree to use and be able to take effective contraceptive birth control measures (Pearl Index < 1) or agree to practice complete abstinence from heterosexual intercourse during the course of the study and for at least 3 months after last application of program treatment. A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 years, or unless she is surgically sterile. Males must agree not to father a child (including not donating sperm) during the course of the trial and for at least 6 months after last administration of study drugs; （11） Previous treatment with combination drug tegafur, gimeracil, and oteracil potassium with seven days before enrollment; （12） Current treatment with Sorivudine; （13） Severe fatigue or bone marrow depression after prior radiotherapy or antineoplastic therapy; （14）There are serious concomitant diseases, such as diabetes mellitus and can not be well controlled by hypoglycemic drugs, clinically serious (that is, active) heart disease, renal failure, liver failure, uncontrolled epilepsy, central nervous system disease or history of mental disorders, hemorrhagic peptic ulcer, intestinal paralysis, intestinal obstruction, etc.; （15） History of other malignancy with a disease-free interval <5 years (Registration is permitted if it has minimal impact on prognosis, such as carcinoma in situ and papillary thyroid cancer); （16） History or current eveidence of brain metastasis; （17）Patients deemed unsuitable for this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of histologically or cytologically confirmed cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-05 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | from the date of enrollment to the earlier of the date of confirmed progression or death from any cause. (assessed up to 12 months
  Progression-free survival is the time from the date of enrollment to the earlier of the date of confirmed progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | from the date of enrollment to death from any cause. (assessed up to 12 months）
  Overall survival is the time from the date of enrollment to death from any cause
Response rates determined by the investigator according to the RECIST(Response Evaluation Criteria in Solid Tumors) v1.1 | Time Frame: from the date of enrollment to end of treatment. (assessed up to 12 months）
  The response rate is the proportion of eligible patients with measurable lesions with a overall response of CR(Complete Response) or PR(Partial Response)
EORTC-QLQ (European Organization for Research and Treatment of Cancer - Quality of life Questionnaire) C30 (version 3.0) | from the date of Screening to end of treatment. (assessed up to 12 months)
  EORTC-QLQ C-30 questionnaires will be performed at screening visit, at pre-dose (Cycle 1 Day1) of every subsequent cycle, at the end of treatment visit. It is a 30-item questionnaire. It has 4-point scales for the item number 1 to 28. These are coded with the same response categories as items 1 to 28, namely "not at all=1" "a little=2" "quite a bit=3" and "very much=4" It has 7-point scale for question number 29 to 30. These are coded with the same response categories as items 29 to 30, namely "worst=1" to "best=7" Total score will be minimum 30 and maximum 126.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No